CLINICAL TRIAL: NCT00337766
Title: Efficacy of Desmopressin (1-deamin0-8-D-arginine-vasopressin) in Reducing Active Microvascular Bleeding After Cardiac Surgery
Brief Title: Desmopressin in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DS/URC/ER/mm 151/DG
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2013-05

CONDITIONS: Hemorrhage; Blood Loss, Surgical; Postoperative Hemorrhage
Keywords: Blood Loss; Postoperative Blood loss
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Desmopressin (DDAVP) (Active Comparator)
  Interventions: Drug: Desmopressin (DDAVP)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin (DDAVP)
  Arms: Desmopressin (DDAVP)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patients undergoing cardiac surgery could develop excessive perioperative bleeding requiring transfusions of blood products.

Desmopressin (DDAVP), already used for patients with von Willebrand syndrome, could reduce bleeding and transfusion requirements in these patients when administered ev (0.3 mg/kg) in 20-30 minutes postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* undergoing cardiac surgery
* excessive bleeding

Exclusion Criteria:

* age<18 y
* not signing written consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Reduce transfusions

SECONDARY OUTCOMES:
Reduced bleeding
Reduce time on mechanical ventilation
Reduced ICU and Hospital stay
Reduced mortality

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Landoni, MD, Study Director — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia.; Giuseppe Crescenzi, MD, Principal Investigator — Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia.
Locations (4):
- Italy (4):
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Università Vita-Salute San Raffaele, Milano, Italia e Istituto Scientifico San Raffaele, Milano, Italia, Milan
  - Istituto Policlinico S.Donato, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa

REFERENCES:
- [Background] Crescenzi G, Landoni G, Biondi-Zoccai G, Pappalardo F, Nuzzi M, Bignami E, Fochi O, Maj G, Calabro MG, Ranucci M, Zangrillo A. Desmopressin reduces transfusion needs after surgery: a meta-analysis of randomized clinical trials. Anesthesiology. 2008 Dec;109(6):1063-76. doi: 10.1097/ALN.0b013e31818db18b. PMID 19034103